CLINICAL TRIAL: NCT01031550
Title: Isoflurane Induced Anesthetic Preconditioning in Elective Liver Resection
Brief Title: Isoflurane Preconditioning for Liver Resections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We no longer had an appropriate patient population.Study closed
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Yuriy Gubenko, MD, Investigator Intiated Dept of Anesthesia, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120090226
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Liver Disease
Keywords: liver resection for liver disease
MeSH Terms: conditions — Liver Diseases | interventions — Isoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard anesthetic management (Active Comparator): standard anesthetic management with propofol 100-150mcg/kg/min
  Interventions: Drug: propofol
- preconditioning with 2 MAC isoflurane group (Experimental): After induction, anesthesia will be maintained with 1MAC (minimum alveolar concentration) of Isoflurane according to age and end-expiratory concentration. Thirty minutes before the anticipated inflow occlusion and commencement of liver transaction, Isoflurane concentration will be gradually increased to 2 MAC over a period of 5 minutes (induction) and maintained at 2 MAC for 10 minutes (preconditioning). Then the concentration of Isoflurane will be decreased to 1 MAC during next 15 minutes (washout).
  Interventions: Drug: isoflurane

INTERVENTIONS:
Drug: isoflurane — isoflurane an anesthetic gas agent administered at specific times at a flow of 2 MAC
  Arms: preconditioning with 2 MAC isoflurane group
Drug: propofol — standard of care
  Other Names: diprivan
  Arms: standard anesthetic management

SUMMARY:
The objective is to examine the efficacy of isoflurane (inhaled anesthetic gas) to induce clinically effective preconditioning in patients undergoing elective hepatic surgery.

DETAILED DESCRIPTION:
Elective liver resection is performed primarily for the treatment of benign and malignant liver tumors1. In addition, with the increasing use of living donor liver transplantation to supplement the inadequate pool of cadaveric organs available, liver resection is performed also in live liver donors2.

Postoperative complications are common following liver resections. Occurrence of complications increases ICU and hospital stay, and resource utilization. The most serious postoperative complication after a liver resection is post-resectional liver failure (PLF)3. Risk factors for the development of PLF are preexisting liver disease, especially cirrhosis, excessive blood loss during liver resection, and liver ischemia and reperfusion injury4-5. Several strategies have been developed to combat excessive intra-operative blood loss including: lowering the central venous pressure6, hypoventilation7, and hepatic inflow occlusion using an atraumatic clamp8 (Pringle's maneuver)9; While inflow occlusion is the most important of these steps, hepatic ischemia and reperfusion is an important sequel to the inflow occlusion. Therefore, interventions which decrease hepatic ischemia reperfusion injury to the liver have the potential to improve outcomes following liver resection.

A strategy that directly modulates the hepatic response to ischemia is ischemic preconditioning (IPC). Classically, IPC has been induced by exposing an organ to brief periods of ischemia and reperfusion before exposing the organ to a more prolonged ischemic insult. In patients undergoing liver resection, IPC decreases postoperative aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels15. IPC is also associated with decreased histological evidence of apoptosis as well as immunohistochemical evidence of increased protective gene expression16 in the liver.

The primary disadvantage of IPC is the direct stress to the target organ as well as the mechanical trauma to major vasculature.

More recently, it has been found that inhaled volatile anesthetics such as Desflurane, Sevoflurane and Isoflurane induce similar preconditioning effects19 without causing any significant direct organ damage. While several animal studies exist, which demonstrate the hepatoprotective effect of volatile anesthetics on the liver23, there is only limited clinical data examining their effect in humans. One recent small clinical study, examining the preconditioning effect of volatile anesthetic on patients undergoing liver surgery, showed that anesthetic pre conditioning (APC) using Sevoflurane significantly decreased the several measures of liver dysfunction postoperatively24.

However, Sevoflurane is partially metabolized by the liver and may increase plasma fluoride concentration. Also, it may react with CO2 absorbent and can produce Compound-A, which in turn has been linked to nephrotoxicity. On the other hand, isoflurane, another inhalational anesthetic agent commonly used during liver surgery also has been shown to have a preconditioning effect in experimental animals, and does not carry the potential side effects of sevoflurane.

Therefore, the primary objective of this study is to examine the efficacy of isoflurane to induce clinically effective preconditioning in patients undergoing elective hepatic surgery.

Study Design:

In this prospective study, patients undergoing elective liver resection with inflow occlusion (Pringle maneuver) at UH, Newark will be randomized (1:1) to either standard anesthetic management with Propofol (No APC group) or anesthetic preconditioning with 2 minimum alveolar concentration (MAC) of isoflurane (APC group). Because preexisting liver disease, especially cirrhosis, is an important determinant of post operative outcomes, and to balance the randomization of subjects regarding this important variable randomization will be stratified into those with and without preexisting liver disease. The primary endpoint is the occurrence of postoperative complications grade IIIb or greater (Clavien's classification). The secondary endpoints are peak postoperative aspartate and alanine aminotransferase (AST and ALT) and total bilirubin (T Bili), length of ICU and hospital stay, and a decrease in liver lipid peroxidation and apoptosis

ELIGIBILITY:
Inclusion Criteria:

* patients with liver tumors undergoing liver resection of > 1 segment liver resection must be performed with inflow occlusion > 30 min

Exclusion Criteria:

* patients undergoing liver resection of one segment or less
* patients undergoing laparoscopic liver resection
* patients in whom the liver resection is performed with no inflow occlusion or inflow occlusion of < 30 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Gubenko, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ-University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be randomized in two strata, those with and without preexisting liver disease. Subjects will be screened in pre admission testing
Pre-assignment Details: Subjects may withdraw consent
Groups:
- Standard Anesthetic Management: standard anesthetic management propofol 100-150mcg/kg/min
- Preconditioning With 2 MAC Isoflurane Group: preconditioning with isoflurane, anesthesia will be maintained with 1MAC of Isoflurane according to age and end-expiratory concentration. Thirty minutes before the anticipated inflow occlusion and commencement of liver transaction, Isoflurane concentration will be gradually increased to 2 MAC over a period of 5 minutes (induction) and maintained at 2 MAC for 10 minutes (preconditioning). Then the concentration of Isoflurane will be decreased to 1 MAC during next 15 minutes (washout).
Period: Overall Study
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Preconditioning With 2 MAC Isoflurane Group: preconditioning with isoflurane anesthesia will be maintained with 1MAC of Isoflurane according to age and end-expiratory concentration. Thirty minutes before the anticipated inflow occlusion and commencement of liver transaction, Isoflurane concentration will be gradually increased to 2 MAC over a period of 5 minutes (induction) and maintained at 2 MAC for 10 minutes (preconditioning). Then the concentration of Isoflurane will be decreased to 1 MAC during next 15 minutes (washout).
- Total: Total of all reporting groups
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 38 (8) | 39 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Complications Grade IIIb or Greater According to Clavien's Classification Which is a Classification System Used to Grade Surgical Complications
Description: Post operative complications grade IIIB or greater according to Clavien's classification: IIIb=complication necessitating an intervention under general anesthesia; Grade IV=Life threatening complications requiring ICU management, IV a =single organ dysfunction, IVb=multi-organ dysfunction; V=death Suffix d(disability)=subject suffers from complication at time of discharge. This label indicates the need for a follow up to fully evaluate the complication.
Time Frame: first 7 post operative days
Population: Due to termination of the study no data analysis was performed.
Groups:
- Preconditioning With 2 MAC Isoflurane Group: preconditioning with isoflurane , anesthesia will be maintained with 1MAC of Isoflurane according to age and end-expiratory concentration. Thirty minutes before the anticipated inflow occlusion and commencement of liver transaction, Isoflurane concentration will be gradually increased to 2 MAC over a period of 5 minutes (induction) and maintained at 2 MAC for 10 minutes (preconditioning). Then the concentration of Isoflurane will be decreased to 1 MAC during next 15 minutes (washout).
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Peak Postoperative AST, ALT and T Bili
Time Frame: first 7 post operative days
Population: Due to termination of the study no data analysis was performed.
Groups:
- Standard Anesthetic Management: standard anesthetic management
- Preconditioning With 2 MAC Isoflurane Group: preconditioning with isoflurane
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Length of ICU and Hospital Stay
Time Frame: first 7 post operative days
Population: Due to termination of the study no data analysis was performed.
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Decrease in Liver Lipid Peroxidation and Apoptosis
Time Frame: first 7 post operative days
Population: Due to termination of the study no data analysis was performed.
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of surgery and 7 days later
Arm/Group | Standard Anesthetic Management | Preconditioning With 2 MAC Isoflurane Group
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

LIMITATIONS AND CAVEATS:
Due to termination of the study no data analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No